CLINICAL TRIAL: NCT02738476
Title: Investigation of the Clinical Outcomes of Patellofemoral Arthroplasty Implanted With the MAKOplasty Knee Resurfacing System in Younger Active Patients
Brief Title: Outcomes of MAKOplasty Patellofemoral Arthroplasty in Younger Active Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cincinnati Sportsmedicine Research and Education Foundation (Other)
Responsible Party: Principal Investigator, Sue Barber-Westin, Director Clinical Studies, Cincinnati Sportsmedicine Research and Education Foundation
Other Study IDs: MAKOplasty PFA-001
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Patellofemoral arthroplasty

SUMMARY:
The primary purpose of this investigation is to report the short-term clinical outcomes (2-3 years) of patellofemoral arthroplasty implanted using the MAKOplasty knee resurfacing system.

DETAILED DESCRIPTION:
The primary purpose of this investigation is to report the short-term clinical outcomes of patellofemoral arthroplasty implanted using the MAKOplasty knee resurfacing system.

The secondary purpose is to compare the short-term outcomes, complication rates, and survival rates of this operation to those of our historical controls of patients who underwent either osteochondral autograft transfer or autologous chondrocyte implantation for full-thickness patellofemoral articular cartilage lesions. The investigators believe these data will provide strong evidence to improve the selection criteria for patellofemoral arthroplasty.

All patients will complete validated questionnaires from the Cincinnati Knee Rating System, including the Sports Activity and Function Form, the Occupational Rating Form, and the Symptom Rating Form. Patients will also complete the SF-12 general health questionnaire. In addition to the above mentioned rating systems, patients will also complete questionnaires on post-surgical expectations and general fitness level.

ELIGIBILITY:
Inclusion Criteria:

* Arthroscopically demonstrated localized and isolated full-thickness articular cartilage lesions (Grade 2B or 3A-B as defined by Noyes & Stabler9) on the patellofemoral joint.
* Lesion is symptomatic as defined by pain, swelling, locking, or catching that affects daily activities.
* Patient provides informed consent.
* Patient agrees to comply with postoperative rehabilitation program.

Exclusion Criteria:

* Obesity (body mass index greater than 35).
* Arthroscopically demonstrated full-thickness articular cartilage lesions (Grade 2B or 3A-B) in the other compartments of the knee.
* Uncorrected varus or valgus malalignment
* Uncorrected knee joint instability
* Knee arthrofibrosis
* Patient unwilling to comply with postoperative rehabilitation
* Significant muscular atrophy and weakness that does not respond to rehabilitation
* History of alcohol or drug abuse within 3 years of the operation.
* Disabling or widespread osteoarthritis or other joint disease in any other joint.
* Presence of a significant connective tissue disease, autoimmune disease, HIV-positive, or immune deficiency syndrome.
* Any contraindications to surgery or other medical disorder that in the opinion of the principal investigator would interfere with the conduct of the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will include 60 patients (men and women) who undergo patellofemoral arthroplasty by one surgeon.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Short-term clinical outcomes of patellofemoral arthroplasty | 3 years
  The clinical outcomes will be determined by comparing the preoperative questionnaire data collected with the 2 and 3-year follow-up data.

SECONDARY OUTCOMES:
Comparison clinical outcomes of patellofemoral arthroplasty with historical controls | 3 years
  The clinical outcomes of patellofemoral arthroplasty will be compared with those of osteochondral autograft transfer and autologous chondrocyte implantation procedures
Comparison of complications, reoperation, and failures rates of patellofemoral arthroplasty with historical controls | 3 years
  The complications, reoperation rates, and failure rates of patellofemoral arthroplasty patients will be compared with those of osteochondral autograft transfer and autologous chondrocyte implantation patients

CONTACTS AND LOCATIONS:
Overall Officials: Frank R Noyes, MD, Principal Investigator — Cincinnati Sportsmedicine and Orthopaedic Center
Locations (1):
- Cincinnati Sportsmedicine and Orthopaedic Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Noyes FR, Fleckenstein CM, Nolan J. Return to Sports in Patients Aged 50 Years or Younger After Robotic-Assisted Patellofemoral Arthroplasty: A 10-Year Experience Reporting High Clinical Benefits and High Patient Satisfaction With Return to an Active Lifestyle. Am J Sports Med. 2024 May;52(6):1514-1526. doi: 10.1177/03635465241237460. Epub 2024 Apr 24. PMID 38656145